CLINICAL TRIAL: NCT03450421
Title: A Randomized, Controlled, Multi-Center Study to Assess the Safety and Efficacy of Actamax™ Adhesion Barrier in Women Undergoing Laparoscopic Abdominopelvic Surgery With a Myomectomy Followed by Second Look Laparoscopy (SLL)
Brief Title: Safety and Efficacy of Actamax™Adhesion Barrier in Women Undergoing Laparoscopic Abdominopelvic Surgery/Myomectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Actamax Surgical Materials LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABS-03UE-2014
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Actamax™Adhesion Barrier (Experimental): Following Myomectomy, subjects randomized to the Actamax™Adhesion Barrier Arm will have up to 30mL of product applied to all sites of surgery (area of treatment/trauma).
  Interventions: Device: Actamax™Adhesion Barrier
- Surgical Control (No Intervention): Myomectomy will be performed with no adhesion barrier application.

INTERVENTIONS:
Device: Actamax™Adhesion Barrier — Actamax™Adhesion Barrier is a degradable hydrogel to be sprayed directly on surgically traumatized tissue. The aim of using the Actamax™ Adhesion Barrier (AB) in this way is to allow damaged and apposing tissue surfaces the opportunity to heal separately without becoming abnormally attached.
  Arms: Actamax™Adhesion Barrier

SUMMARY:
Women undergoing laparoscopic abdominopelvic surgery with a planned, second look laparoscopy within 8-12 (+4) weeks will be enrolled. All subjects must undergo myomectomy with/without treatment of co-existing pathology e.g. (+/-) adhesions and/or (+/-) endometriosis, and/or (+/-) adenomyosis, and/or (+/-) ovarian cyst(s). The value of the second look laparoscopy (SLL) must be confirmed by the investigator to be of clinical benefit to the subject. The subject must be desirous of future fertility and willing to undergo the SLL to assess whether pathology (e.g. adnexal adhesions or endometriosis) exists which could be treated with a goal of improving their likelihood of conceiving and progressing to full term.

ELIGIBILITY:
Preoperative Inclusion Criteria:

* Understand and be able to follow the requirements of the protocol including personally signing and dating an IRB approved Informed Consent Form prior to undergoing any protocol related procedures,
* Be a premenopausal female, > 18 and < 44 years old,
* Be thought to have uterine fibroids requiring laparoscopic abdominopelvic surgery that will require a > 3 cm posterior uterine incision (including repeat myomectomy/previous uterine artery embolization for fibroid), and/or +/- adhesions, and/or +/- endometriosis, and/or +/- adenomyosis and/or ovarian cyst(s),
* Wish to retain her fertility and be considered to clinically benefit from a SLL, in the investigator's opinion,
* Have a willingness to undergo a second look laparoscopy if surgeon considers it clinically beneficial to the subject,
* Have a negative pregnancy test within 5 days of surgery,
* Agree to avoid pregnancy using adequate forms of contraception (oral contraceptive pill, condom, no sexual intercourse), and is aware and agrees to avoid pregnancy for a minimum of 12 weeks or to SLL (whichever is greater) to allow for healing of the uterine scar following myomectomy,
* Is willing, able and likely to fully comply with study procedures and restrictions including follow-up,
* Be in good health including an ASA (American Society of Anesthesiologists) score of 2 or less,
* Have undergone a satisfactory physical and medical assessment with no clinically significant and relevant abnormalities.

Intraoperative Inclusion Criteria:

* The subject underwent a laparoscopic myomectomy with at least (1) posterior uterine serosal incision of > 3 cm in length,
* The subject meets all intraoperative inclusion/exclusion criteria prior to randomization,

And

• At the completion of the procedure, before randomization, the surgeon believes that the subject will clinically benefit from a second look laparoscopy to preserve fertility.

Preoperative Exclusion Criteria:

* Are unable to give their own written informed consent,
* Have completed her family planning with no desire to maintain fertility,
* Are considered to have no potential clinical benefit from a second look laparoscopy,
* Are currently pregnant (including ectopic pregnancy),
* Are breastfeeding,
* Are within 6 weeks post-partum,
* Have received or are expected to receive another anti-adhesive treatment within 30 days prior to enrollment or during enrollment up to adhesion evaluation at second look laparoscopy,
* Are currently or have been enrolled within the last 30 days in another interventional study.
* Have received or are expected to receive any other investigational product or technique within 30 days prior to or during enrollment,
* Have had cancer within 5 years of the initial surgery with the exception of basal cell carcinoma,
* Have known allergy to dextran, PEG, or FD&C Blue #1,
* Have had bilateral salpingectomy,
* Have had a hysterectomy,
* Are scheduled to undergo concomitant non-gynecologic surgery,
* Have pre-operative imaging results with:
* Largest fibroid diameter < 2 cm, or
* Largest intramural fibroid diameter >10 cm, or
* More than 5 intramural fibroids with a diameter of > 8 cm, and/or
* Adenomyoma >10 cm.
* Have a history where it is expected that complete adhesiolysis will be impossible,
* Have clinically significant abnormal blood results,
* Have clinically relevant hemochromatosis, hepatic, renal, autoimmune, lymphatic, hematological or coagulation disorders,
* Have insulin dependent diabetes mellitus,
* Are receiving concurrent systemic corticosteroids, antineoplastic agents and/or radiation therapy,
* Have had previous abdominal or pelvic radiation therapy,
* Have active pelvic or abdominal infection, or other active infection with fever >100°F/38°C,
* Have a known history of methicillin-resistant Staphylococcus aureus (MRSA), HIV, HBV or HCV.

Intraoperative Exclusion Criteria:

* Have cancer detected at surgery,
* Are pregnant, including ectopic pregnancy,
* Have a non-gynecologic surgical procedure or entry into the bowel, bladder, or ureter,
* Have a hysterectomy or other gynecologic procedure that would render the subject unable to conceive,
* Have incomplete lysis of any pre-existing pathological adhesions,
* Have extensive enterolysis,
* Have incomplete surgical treatment of endometriosis,
* Receive the administration of a product that will interfere with the application of Actamax™ Adhesion Barrier,
* Receive the use of an approved or unapproved product or strategy for the purpose of preventing adhesion development,
* Receive fibrin glue, surgical sealant, or other hemostatic agent,
* Undergo an open procedure (other than mini laparotomy to remove fibroids),
* Undergo a posterior colpotomy,
* Undergo insufflation with a gas other than CO2,
* Undergo Laprolift or similar device for elevation of the abdominal wall, as an alternative to CO2 insufflation,
* Undergo abdominal cavity heating, humidification or oxygenation,
* Receive irrigants containing, glucocorticoids, antihistamines, heparin or antiseptic additives,
* Have any instillates left at the end of surgery,
* Have a postoperative drain,
* Undergo laparoscopic myomectomy without at least one posterior uterine serosal incision of > 3 cm in length,
* Undergo a diagnostic hysteroscopy or polypectomy or therapeutic hysteroscopy which includes any of the following:

  1. Undertaken during or following the laparoscopic myomectomy,
  2. Treatment of fibroids >3 cm,
  3. Solution other than Lactated Ringer's Solution (LRS) used for uterine distention,
  4. Laparoscopic filming commenced after removal of LRS.
* If, in the opinion of the surgeon, subject would have no clinical benefit for a SLL.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Adhesion Free at Sites of Surgery at SLL | 8-12 weeks postoperatively but out to 16 weeks where circumstances require (vacations, etc.)
  The primary efficacy outcome measure will be being adhesion free at sites of surgery throughout the whole abdominopelvic cavity at SLL.

CONTACTS AND LOCATIONS:
Overall Officials: Trudy Estridge, Study Director — Actamax Surgical Materials LLC